CLINICAL TRIAL: NCT05609851
Title: The Relationship of Physical Performance With Perceived Occupational Competence and Value in Elderly
Brief Title: Relationship Occupation and Physical Performance in Elderly
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Ogr Uyesi Tuba MADEN, Assisstanf Profesor, University of Gaziantep
Other Study IDs: 2020/280
Record Dates: First submitted 2022-10-28; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Old Age; Atrophy; Elderly; Occupational Balance; Postural Balance; Physical Performance
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: A physical performance test will be applied to the group and Questionnaires related to occupation will be made to individuals.
  Interventions: Other: Short Physical Performance Batary; Other: Occupational Balance Self-Assessment

INTERVENTIONS:
Other: Short Physical Performance Batary — The SPPB includes usual walking speed over 4 m, five chair-stands test, and balance test. A score (scale: 0-4) was assigned to performance on time to rise five times from a seated position, standing balance, and 4-m walking velocity. Individuals received a score of 0 for each task they were unable to complete. Participants coded in the "unable to perform" category included (a) those who tried but were unable and (b) the interviewer or participant felt it was unsafe. Summing the three individual categorical scores, a summary performance score was created for each participant (range: 0-12), with higher scores indicating better lower body function.
Other: Occupational Balance Self-Assessment — The Occupational Self-Assessment (OSA) is a self-reported assessment tool consisting of 21 items in which the patient rates their occupational competence (i.e., how well they do) and value (i.e., how important it is to them). The first 11 items are related to skills and occupational performance, the next five items concern habitation (including habits and roles), and the last five items correspond to volition (including personal causation, values, and interests). In the OSA, each item is scored on two separate 4-point scales, one for occupational competence (1 = I have a lot of problems doing this; 4 = I do this extremely well) and the other for value (1 = This is not important to me; 4 = This is most important to me).
  The individual item scores are summed to obtain separate total scores for competence and value. Higher total scores indicate higher occupational competence and value.

SUMMARY:
Occupational competence indicates participating in a variety of occupations to meet the standards expected of the individuals' valued roles to sustain a pattern of occupational attitudes that is significant and satisfying. Physical performance declines with age. This causes problems with balance and falling. Balance and falling losses can also affect occupation. Our study was conducted to examine the relationship between physical performance and occupational balance in elderly individuals. According to the power analysis, it is planned to include the individual in the study. Individuals will only be evaluated and the relationship between scale results will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 65 and over will be included.

Exclusion Criteria:

* Having visual-hearing loss that prevents them from making evaluations,
* Individuals with poor co-operation will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Volunteers aged 65 and over older adults.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OSA | through study completion, an average of one month
  The Occupational Self-Assessment (OSA) is a self-reported assessment tool consisting of 21 items in which the patient rates their occupational competence (i.e., how well they do) and value (i.e., how important it is to them). The first 11 items are related to skills and occupational performance, the next five items concern habitation (including habits and roles), and the last five items correspond to volition (including personal causation, values, and interests). In the OSA, each item is scored on two separate 4-point scales, one for occupational competence (1 = I have a lot of problems doing this; 4 = I do this extremely well) and the other for value (1 = This is not important to me; 4 = This is most important to me).
  The individual item scores are summed to obtain separate total scores for competence and value. Higher total scores indicate higher occupational competence and value.

CONTACTS AND LOCATIONS:
Overall Officials: tuba maden, PhD, Principal Investigator — University of Gaziantep
Locations (1):
- Tuba Maden, Gaziantep, Turkey (Türkiye)